CLINICAL TRIAL: NCT02057627
Title: Dyadic Intervention for Women at Risk for Postpartum Depression and Their Infants
Brief Title: Mother-Infant Intervention for Postpartum Depression and Associated Mother-Infant Relationship Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Janice H. Goodman, Associate Professor, Spaulding Rehabilitation Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R21HD065156-01 (NIH)
Record Dates: First submitted 2014-02-05; First posted 2014-02-07 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Perinatal Dyadic Psychotherapy (Experimental): The Perinatal Dyadic Psychotherapy intervention consists of 8 home-based, nurse-delivered mother-infant sessions consisting of (a) a supportive, relationship-based, mother-infant psychotherapeutic component, and (b) a developmentally based infant-oriented component focused on promoting positive mother-infant interactions. The 8 sessions take place over three months with weekly 4 sessions (weeks 1 through 4) followed by 4 every other week sessions (weeks 5 through 8)
  Interventions: Behavioral: Perinatal Dyadic Psychotherapy
- Standard care plus depression monitoring (Placebo Comparator): Standard care plus depression monitoring by phone on a schedule comparable to the intervention groups' home visits. Eight phone calls will take place over three months with weekly 4 calls (weeks 1 through 4) followed by 4 every other week calls (weeks 5 through 8). Phone monitoring will include administration of the Edinburgh Postnatal Depression Scale.
  Interventions: Behavioral: Placebo Comparator

INTERVENTIONS:
Behavioral: Perinatal Dyadic Psychotherapy — 8-session mother-infant psychotherapy (Perinatal Dyadic Psychotherapy) delivered by nurse-interventionists in participant's homes over 3 months
  Arms: Perinatal Dyadic Psychotherapy
Behavioral: Placebo Comparator — Standard care plus depression monitoring by phone
  Arms: Standard care plus depression monitoring

SUMMARY:
Maternal depression and mother-infant relationship dysfunction have reciprocal effects on each other. An integrated approach addressing both problems simultaneously may improve outcomes. Perinatal Dyadic Psychotherapy (PDP) was developed to prevent/decrease postpartum depression and facilitate optimal mother-infant relationships. The purpose of this pilot study is to determine the feasibility, acceptability, and preliminary efficacy of PDP. Depressed first-time mothers (meeting diagnostic criteria for depression and/or with high depression symptom levels) and their 6-week-old infants will be randomized to receive either the PDP intervention or a control condition. The PDP intervention consists of 8 home-based, nurse-delivered mother-infant sessions consisting of (a) a supportive, relationship-based, mother-infant psychotherapeutic component, and (b) a developmentally based infant-oriented component focused on promoting positive mother-infant interactions. Control mothers will receive usual care plus depression monitoring by phone. Data will be collected at baseline, post-intervention, and 3 month follow-up. Assessments included maternal depression (diagnosis and severity), maternal anxiety (diagnosis and severity), parenting stress, and mother-infant interaction.

ELIGIBILITY:
Inclusion Criteria:

* First-time, English-speaking mothers of healthy singleton newborns
* Positive screen (> 10) on Edinburgh Postnatal Depression Scale

Exclusion Criteria:

* Suicidal ideation
* Currently receiving depression treatment
* Meets criteria for bipolar disorder and/or lifetime or current psychotic disorder

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline on maternal depression diagnosis immediately following the 3 month intervention and at 3 months post-intervention as measured by the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID) | baseline, 3 months (post-intervention) and 6 months (follow-up)
Change from baseline in maternal depressive symptom scores immediately following the 3 month intervention and at 3 months post-intervention as measured by the Edinburgh Postnatal Depression Scale | baseline, 3 months (post-intervention) and 6 months (follow-up)
Mother-infant interaction (videotaped and coded) immediately following the 3 month intervention and at 3 months post-intervention | 3 months (post-intervention) and 6 months (follow-up)

SECONDARY OUTCOMES:
Change from baseline in maternal anxiety diagnosis immediately following the 3 month intervention and at 3 months post-intervention per Structured Clinical Interview for DSM-IV Axis I Disorders (SCID) | baseline, 3 months (post-intervention) and 6 months (follow-up)
Maternal parenting stress immediately following the 3 month intervention and at 3 months post-intervention as measured by the Parenting Stress Index - Short Form (PSI-SF) | 3 months (post-intervention) and 6 months (follow-up)
Change from baseline in maternal anxiety symptom level immediately following the 3 month intervention and at 3 months post-intervention as measured by the State-Trait Anxiety Inventory - State (STAI-State) | baseline, 3 months (post-intervention), 6 months (follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Janice H Goodman, PhD, Principal Investigator — MGH Institute of Health Professions
Locations (1):
- MGH Insiitute of Health Professions, Boston, Massachusetts, United States

REFERENCES:
- [Result] Goodman JH, Guarino AJ, Prager JE. Perinatal dyadic psychotherapy: design, implementation, and acceptability. J Fam Nurs. 2013 Aug;19(3):295-323. doi: 10.1177/1074840713484822. Epub 2013 Apr 5. PMID 23562990